CLINICAL TRIAL: NCT02641652
Title: A Randomized Controlled Trial of Sertraline in Paroxysmal Arterial Hypertension (ATRAX Trial)
Brief Title: A Randomized Controlled Trial of Sertraline in Paroxysmal Arterial Hypertension
Acronym: ATRAX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Olomouc (Other)
Collaborators: Brno University Hospital (Other); St. Anne (Unknown); University Hospital Ostrava (Other); Tomas Bata Hospital, Czech Republic (Other); Prerov Hospital (Unknown); Valasske Mezirici Hospital (Unknown); Thomayer University Hospital (Other); Vsetin Hospital (Unknown)
Responsible Party: Principal Investigator, Jan Vaclavík, Jan Václavík, MD. Ph.D. Assoc. Prof., Palacky University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRAX
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: paroxysmal hypertension; pseudopheochromocytoma
MeSH Terms: conditions — Hypertension | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sertraline (Active Comparator): sertraline, 25 mg once daily for first 7 days, then 50 mg once daily for the rest of the trial
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — 25 mg once daily for first 7 days, then 50 mg once daily for the rest of the trial
  Arms: Sertraline
Drug: Placebo — 1/2 tablet once daily for first 7 days, then 1 tablet once daily for the rest of the trial
  Arms: Placebo

SUMMARY:
There is currently no established treatment for paroxysmal hypertension, but selective serotonin reuptake inhibitors showed good effect in previous reports. This double-blind, placebo controlled, prospective multicenter clinical trial will assess the efficacy of sertraline on cessation or reduction of symptoms of paroxysmal arterial hypertension. 136 patients with documented hypertensive paroxysms with abrupt elevations of blood pressure and distressful physical symptoms will be randomized in a 1:1 ratio to receive sertraline, 50 mg daily, or matching placebo as an add-on to their chronic medication. Effect of the treatment on patient symptoms, office and ambulatory blood pressure and side effects will be evaluated after 3 months. If proven effective, sertraline might become a standard treatment for this condition.

ELIGIBILITY:
Inclusion Criteria:

Study will enroll adult patients (age >18 years) with hypertensive paroxysms during the past 6 months (preferably during the past 6 weeks) - abrupt elevations of systolic blood pressure (BP) ≥20% compared to previous measured systolic BP value before paroxysm, or ≥20% compared to mean systolic BP on 24-hour ambulatory blood pressure monitoring (ABPM), or ≥20% compared to measured office systolic BP, documented by a clinician or home blood pressure monitor, requiring physician or emergency room visit or the use of any rescue antihypertensive medication. Hypertensive paroxysms may be accompanied by abrupt onset of one or more distressful physical symptoms, such as headache, chest pain, dizziness, nausea, palpitations, flushing, and diaphoresis.

Exclusion Criteria:

Pregnancy or breastfeeding, hypersensitivity to sertraline (Zoloft®) or of the the components of this drug. Current use of sertraline or any other selective serotonin reuptake inhibitor (SSRI), mono-amin oxidase (MAO) inhibitors, selegiline, moclobemide, linezolide, pimozide. Current use of other serotoninergic drugs (eg. tryptofane, triptane and other 5-HT agonists), tramadol or dopamine antagonists (including antipsychotics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
difference in the rate of paroxysmal hypertension symptoms cessation between sertraline and placebo groups | 3 months of treatment
difference in the rate of paroxysmal hypertension symptoms reduction between sertraline and placebo groups | 3 months

SECONDARY OUTCOMES:
difference in the fall of mean office and ambulatory systolic and diastolic blood pressure between groups | 3 months
side effects of the treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vaclavik, MD. Ph.D. Assoc. Prof, Study Chair — University Hospital Olomouc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mann SJ. Severe paroxysmal hypertension (pseudopheochromocytoma): understanding the cause and treatment. Arch Intern Med. 1999 Apr 12;159(7):670-4. doi: 10.1001/archinte.159.7.670. PMID 10218745
- [Background] Eisenhofer G, Sharabi Y, Pacak K. Unexplained symptomatic paroxysmal hypertension in pseudopheochromocytoma: a stress response disorder? Ann N Y Acad Sci. 2008 Dec;1148:469-78. doi: 10.1196/annals.1410.019. PMID 19120143
- [Background] Pickering TG, Clemow L. Paroxysmal hypertension: the role of stress and psychological factors. J Clin Hypertens (Greenwich). 2008 Jul;10(7):575-81. doi: 10.1111/j.1751-7176.2008.07844.x. PMID 18607143
- [Background] Mann SJ. Severe paroxysmal hypertension (pseudopheochromocytoma). Curr Hypertens Rep. 2008 Feb;10(1):12-8. doi: 10.1007/s11906-008-0005-2. PMID 18367021
- See also: University Hospital Olomouc — http://www.fnol.cz
- See also: Faculty of Medicine and Dentistry, Palacký University — http://www.lf.upol.cz/en/